CLINICAL TRIAL: NCT03637101
Title: Ischemia Modified Albumin as a Biomarker for Prediction of Poor Outcome in Patients With Traumatic Brain Injury. Observational Cohort Study
Brief Title: Ischemia Modified Albumin in Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rania Samir Fahmy, Lecturer of Anesthesia, surgical intensive care and pain mangement, Kasr El Aini Hospital
Other Study IDs: N-23-2018
Record Dates: First submitted 2018-08-04; First posted 2018-08-17 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Traumatic Brain Injury
Keywords: Ischemia modified albumin; Traumatic brain injury; Troponin; Conscious Level; Poor outcome
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ischemia modified albumin (IMA) — Ischemia modified albumin is a biomarker for cardiac ischemia and acute stroke whether ischemic or hemorrhagic

SUMMARY:
In the current study the investigators intend to evaluate the role of Ischemia modified albumin (IMA) in the prediction of poor outcome in patients with traumatic brain injury (TBI). The investigators hypothesize that IMA will be elevated in patients with traumatic brain injury due to the excessive production of reactive oxygen species by the injured brain.

DETAILED DESCRIPTION:
Consecutive adult patients who were admitted with TBI, blood samples were taken once written informed consent obtained. Initial evaluation on admission was performed simultaneously by ICU physician and a neurosurgical resident by means of a detailed physical and neurological examination. Demographic characteristics and vascular risk factors (hypertension, diabetes mellitus, hyperlipidemia, and peripheral ischemic disease) were recorded in details. Also, Routine blood tests, including full blood count, coagulation tests, glucose level, renal and hepatic function tests, total protein, and albumin levels; chest radiography were done.

CT scan will be performed in all the cases for the confirmation of TBI. Glasgow coma scale (GCS) was assessed on admission and recorded and assessed daily to evaluate prognosis. Patients were monitored by BP, ECG, and Pulse oximetry. All patients received standard medical treatment which included anti-edema measures mannitol 20%, 0.25-0.5 g/kg over 20 min, (not exceeding a total of 2 g/kg of body weight in 24 h) in patients with symptoms of raised intracranial pressure, and other supportive therapy for the treatment of concurrent illnesses such as hypertension and diabetes mellitus.

Biochemical Assessments:

Blood samples from TBI patients were collected immediately at the time of admission to the ICU and 24 hours later. Samples were centrifuged at 2500 RPM for 15 minutes and obtained serum samples were stored at -20oC.

IMA was measured by the colorimetric method and results were presented in absorbance units (ABSU).

Data collection

* Patients' characteristics: age, gender, BMI, cause of ICU admission.
* IMA will be measured at time of admission to ICU and 24h later
* Other data collections:

  * Hear rate (HR), systolic blood pressure,central venous pressure (CVP), body temperature. All hemodynamic parameters were measured and recorded at time of admission and every 2 hours for 24 hours
  * Length of ICU stay
  * 28-day mortality
  * Troponin I level on admission.
  * GCS at admission and daily till mortality or discharge

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* Patients with isolated head injury

Exclusion Criteria:

* Age < 18 years old
* Pregnant patient
* Acute hepatitis or severe liver disease (Child-Pugh class C)
* Patients with recent pulmonary embolism
* Patients with unstable angina or recent myocardial infarction (MI)
* Peripheral arterial disease
* Acute stroke
* Chronic renal failure (CRF)
* Hypoalbuminemia less than 3.5
* Patients with other organs injury
* Penetrating head injury
* Head trauma more than 24 hours before admission
* Patients with known inflammatory or autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who were admitted to the trauma and neurosurgical ICU with isolated traumatic brain injury
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Correlation between IMA and mortality following TBI | The number of patients who died within 28 days from admission to ICU after TBI and who were investigated for IMA upon admission to ICU
  IMA in ng/ml will be measured at time of admission to ICU and correlated with 28 day mortality

SECONDARY OUTCOMES:
Correlation between 24 hours IMA and mortality following TBI | The number of patients who died within 28 days from admission to ICU after TBI and who were investigated for IMA 24 hours after admission to ICU
  IMA in ng/ml will be measured 24 hours after admission to ICU and correlated with 28 day mortality
The incidence of patients with elevated IMA | IMA on admission to ICU and after 24 hours
  The percentage of patients having elevated IMA in ng/ml from the recruited patients with traumatic brain injuries.
The degree of correlation between severity of TBI and IMA | Glasgow coma scale immediately on admission to the ICU, IMA will be collected on admission to ICU and after 24 hours
  The severity of traumatic brain injury classified by Glasgow Coma Scale as mild 13-15, moderate 9-12 or severe 3-8 and the IMA levels in ng/ml in those patients.
The degree of correlation between mild TBI and ICU length of stay | The number of days in ICU till discharge or mortality up to 28 days post admission
  The number of days spent in ICU for patients with mild TBI (GCS 13-15)
The degree of correlation between moderate TBI and ICU length of stay | The number of days in ICU till discharge or mortality up to 28 days post admission
  The number of days spent in ICU for patients with moderate TBI (GCS 9-12)
The degree of correlation between severe TBI and ICU length of stay | The number of days in ICU till discharge or mortality up to 28 days post admission
  The number of days spent in ICU for patients with severe TBI (GCS 3- 8)
The degree of correlation between severity of TBI and and deterioration of conscious level | Glasgow coma scale immediately on admission to the ICU and daily till mortality or discharge up to 28 days post admission
  The severity of traumatic brain injury classified by Glasgow Coma Scale as mild 13-15, moderate 9-12 or severe 3-8 on admission and the Glasgow coma scale on the following days in the ICU til mortality or discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Aini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nayak AR, Kashyap RS, Kabra D, Purohit HJ, Taori GM, Daginawala HF. Prognostic significance of ischemia-modified albumin in acute ischemic stroke patients: A preliminary study. Ann Neurosci. 2011 Jan;18(1):5-7. doi: 10.5214/ans.0972.7531.1118103. PMID 25205910
- [Background] Sbarouni E, Georgiadou P, Kremastinos DT, Voudris V. Ischemia modified albumin: is this marker of ischemia ready for prime time use? Hellenic J Cardiol. 2008 Jul-Aug;49(4):260-6. No abstract available. PMID 18935713
- [Background] Roy D, Quiles J, Gaze DC, Collinson P, Kaski JC, Baxter GF. Role of reactive oxygen species on the formation of the novel diagnostic marker ischaemia modified albumin. Heart. 2006 Jan;92(1):113-4. doi: 10.1136/hrt.2004.049643. No abstract available. PMID 16365361
- [Background] Chong ZZ, Li F, Maiese K. Oxidative stress in the brain: novel cellular targets that govern survival during neurodegenerative disease. Prog Neurobiol. 2005 Feb;75(3):207-46. doi: 10.1016/j.pneurobio.2005.02.004. Epub 2005 Apr 26. PMID 15882775
- [Background] Riera M, Llompart-Pou JA, Carrillo A, Blanco C. Head injury and inverted Takotsubo cardiomyopathy. J Trauma. 2010 Jan;68(1):E13-5. doi: 10.1097/TA.0b013e3181469d5b. PMID 19065115
- [Background] Prathep S, Sharma D, Hallman M, Joffe A, Krishnamoorthy V, Mackensen GB, Vavilala MS. Preliminary report on cardiac dysfunction after isolated traumatic brain injury. Crit Care Med. 2014 Jan;42(1):142-7. doi: 10.1097/CCM.0b013e318298a890. PMID 23963125
- [Background] Hasanin A, Kamal A, Amin S, Zakaria D, El Sayed R, Mahmoud K, Mukhtar A. Incidence and outcome of cardiac injury in patients with severe head trauma. Scand J Trauma Resusc Emerg Med. 2016 Apr 27;24:58. doi: 10.1186/s13049-016-0246-z. PMID 27121183
- [Background] Myburgh JA, Cooper DJ, Finfer SR, Venkatesh B, Jones D, Higgins A, Bishop N, Higlett T; Australasian Traumatic Brain Injury Study (ATBIS) Investigators for the Australian; New Zealand Intensive Care Society Clinical Trials Group. Epidemiology and 12-month outcomes from traumatic brain injury in australia and new zealand. J Trauma. 2008 Apr;64(4):854-62. doi: 10.1097/TA.0b013e3180340e77. PMID 18404048